CLINICAL TRIAL: NCT00548730
Title: A Clinical Comparison Trial of White Light Bronchoscopy, Autofluorescence Bronchoscopy and Narrow Band Imaged Bronchoscopy
Brief Title: Comparison Trial of White Light, Autofluorescence and Narrow Band Imaging Bronchoscopy
Acronym: NWA
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient enrollment
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Administration Director, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Other Study IDs: MMC07/06VA14
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer
Keywords: Bronchoscopy; Endoscopy; Image Enhancement; Autofluorescence; Narrow Band Image
MeSH Terms: conditions — Lung Neoplasms | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endobronchial biopsies of normal and abnormal mucosa for histopathology
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- White Light Bronchoscopy: Patients with known or suspected malignancies of the lung and with a medical indication for a bronchoscopy will have images taken with white light bronchoscopy
  Interventions: Procedure: Bronchoscopy
- Autofluorescence Bronchoscopy: Patients with known or suspected malignancies of the lung and with a medical indication for a bronchoscopy will have images taken with autofluorescence bronchoscopy
  Interventions: Procedure: Bronchoscopy
- Narrow Band Imaged Bronchoscopy: Patients with known or suspected malignancies of the lung and with a medical indication for a bronchoscopy will have images taken with narrow band imaged bronchoscopy
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — The endoscopic examination of the bronchial tree will be performed using a commercially available flexible fluorescence bronchoscope and the flexible white light video-bronchoscope. Biopsies are taken of a normal region and all abnormal regions.
  Other Names: AF bronchoscope (11004BI); NBI bronchoscope (BF-T180)

SUMMARY:
The purpose of the study is to compare the three methods of bronchoscopic imaging to determine what combination is optimum to identify neoplastic mucosal abnormalities. The ability to decrease the rate of false-positive and false negative findings of bronchoscopy also will be studied for each spectroscopic technique separately and for their combination.

DETAILED DESCRIPTION:
Patients with known or suspected malignancies of the lung and with a medical indication for a bronchoscopy will be invited to participate in the study. All patients must be over 18 years old and must sign informed consent. The endoscopic examination of the bronchial tree will be performed using a commercially available flexible fluorescence bronchoscope (11004BI; Karl Storz; Culver City, CA) and the flexible white light video-bronchoscope (BF-T180; Olympus; Center Valley, PA).

Images obtained will be photographed using both video recordings and parallel images of white light and imaged bronchoscopy. These digital images will be electronically stored and evaluated at a later time. Biopsies will be obtained of all suspected abnormalities. These will be correlated with the images.

Images will be identified as normal, suspect or abnormal based upon each modality independently, paired with the spectral image and all three combined. The control will be an area considered normal by all modes of bronchoscopy. Images will be graded at the time of bronchoscopy. Later, all images will be graded in a blind fashion by two independent bronchoscopists. Standard statistical analysis using paired Student's t test will be applied. We anticipate that the combination of one or more imaged bronchoscopy techniques will increase accuracy by 25%. Power calculation to detect such a difference will require 140 abnormal specimens. If 50% of patients examined have an abnormality, the study population will need to be around 300 patients.

Histopathology reports will be obtained on all specimens. Abnormal results will be discussed with the individual patient and appropriate procedures will be performed based upon best medical practices. These procedures and patient follow-up are beyond the scope of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung abnormalities that have an indication for bronchoscopy

Exclusion Criteria:

* Inability to tolerate bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with known or suspected malignancies of the lung and with a medical indication for a bronchoscopy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-10-01 (Actual); Primary Completion 2009-05-31 (Actual); Study Completion 2009-05-31 (Actual)

PRIMARY OUTCOMES:
Degree of correlation between three different bronchoscopic images | One day

SECONDARY OUTCOMES:
Elimination of false positives and negative bronchoscopic examinations for neoplasia | One day

CONTACTS AND LOCATIONS:
Overall Officials: Joseph LoCicero, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Background] DaCosta RS, Wilson BC, Marcon NE. Light-induced fluorescence endoscopy of the gastrointestinal tract. Gastrointest Endosc Clin N Am. 2000 Jan;10(1):37-69, vi. PMID 10618453
- [Background] Gono K, Obi T, Yamaguchi M, Ohyama N, Machida H, Sano Y, Yoshida S, Hamamoto Y, Endo T. Appearance of enhanced tissue features in narrow-band endoscopic imaging. J Biomed Opt. 2004 May-Jun;9(3):568-77. doi: 10.1117/1.1695563. PMID 15189095
- [Background] Vincent BD, Fraig M, Silvestri GA. A pilot study of narrow-band imaging compared to white light bronchoscopy for evaluation of normal airways and premalignant and malignant airways disease. Chest. 2007 Jun;131(6):1794-9. doi: 10.1378/chest.06-2794. Epub 2007 May 15. PMID 17505042
- [Background] Lee P, Brokx HA, Postmus PE, Sutedja TG. Dual digital video-autofluorescence imaging for detection of pre-neoplastic lesions. Lung Cancer. 2007 Oct;58(1):44-9. doi: 10.1016/j.lungcan.2007.04.009. Epub 2007 May 29. PMID 17532537
- [Background] Ueno K, Kusunoki Y, Imamura F, Yoshimura M, Yamamoto S, Uchida J, Tsukamoto Y. Clinical experience with autofluorescence imaging system in patients with lung cancers and precancerous lesions. Respiration. 2007;74(3):304-8. doi: 10.1159/000093233. Epub 2006 May 5. PMID 16679756
- [Background] Jang TW, Oak CH, Chun BK, Jung MH. Detection of pre-invasive endobronchial tumors with D-light/autofluorescence system. J Korean Med Sci. 2006 Apr;21(2):242-6. doi: 10.3346/jkms.2006.21.2.242. PMID 16614508
- [Background] Haussinger K, Becker H, Stanzel F, Kreuzer A, Schmidt B, Strausz J, Cavaliere S, Herth F, Kohlhaufl M, Muller KM, Huber RM, Pichlmeier U, Bolliger ChT. Autofluorescence bronchoscopy with white light bronchoscopy compared with white light bronchoscopy alone for the detection of precancerous lesions: a European randomised controlled multicentre trial. Thorax. 2005 Jun;60(6):496-503. doi: 10.1136/thx.2005.041475. PMID 15923251